CLINICAL TRIAL: NCT00362336
Title: Immunogenicity Study of a DTaP-IPV-Hep B-PRP~T Combined Vaccine in Comparison to CombAct-HIB® Concomitantly Administered With Engerix B® Paediatric and OPV at 6, 10, and 14 Weeks of Age in South African Infants
Brief Title: Comparison of DTaP-IPV-Hep B-PRP~T Combined Vaccine to CombAct-HIB® Concomitantly Given With Engerix B® Paediatric and OPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L15
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis B; Polio; Diphtheria; Pertussis; Haemophilus Influenzae Type b
Keywords: Hepatitis B; Polio; Diphtheria; Pertussis; H. influenzae type b
MeSH Terms: conditions — Hepatitis B; Poliomyelitis; Diphtheria; Whooping Cough; Haemophilus Infections | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: DTaP-IPV-Hep B-PRP-T (Experimental)
  Interventions: Biological: DTaP-IPV-HB-PRP~T
- Group 2: CombAct-HIB™ + OPV (Experimental)
  Interventions: Biological: CombAct-HIB®
- Group 3: DTaP-IPV-Hep B-PRP-T (ENGERIX B™ at birth) (Active Comparator)
  Interventions: Biological: Engerix B® Pediatric

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T — 0.5 mL, Intramuscular (IM)
  Arms: Group 1: DTaP-IPV-Hep B-PRP-T
Biological: CombAct-HIB® — 0.5 mL, IM
  Arms: Group 2: CombAct-HIB™ + OPV
Biological: Engerix B® Pediatric — 0.5 mL, IM
  Arms: Group 3: DTaP-IPV-Hep B-PRP-T (ENGERIX B™ at birth)

SUMMARY:
The purpose of this study is to document the immunological response to the investigational hexavalent vaccine at the 6, 10, and 14 weeks schedule

The primary objective is to demonstrate that the hexavalent DTaP-IPV-HB-PRP~T combined vaccine does not induce lower immune responses than CombAct-HIB® with Engerix B® Paediatric and OPV in terms of seroprotection rates to Diphtheria (D), Tetanus (T), polio, Hepatitis B (HB), and Polyribosyl ribitol phosphate (PRP), one month after a 3-dose primary series (6, 10, and 14 weeks) with no HB vaccination at birth.

The secondary Objectives are:

To describe the safety in terms of any adverse events in the first 28 days after each injection and any serious adverse events during the entire trial.

To describe Immunogenicity after the primary series and prior to and after a booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 3 day old infants
* Mother seronegative for Human Immunodeficiency Virus (HIV)
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg
* Apgar score >7 at 5 or 10 minutes of life
* Informed consent form signed by a parent or other legal guardian and by an independent witness if the parent or other legal guardian is illiterate
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Current or planned participation in another clinical trial during the entire duration of the present trial
* Suspected congenital or acquired immunodeficiency
* Suspected maternal acute seroconversion syndrome to HIV after 24 weeks gestation based on clinical history
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received since birth
* Any planned vaccination (except Bacille Calmette Guérin and trial vaccinations) from birth to 18 weeks of age
* Oral Poliovirus Vaccine (OPV) administration at birth
* Known maternal history of HIV, Hepatitis B (HB) (HbsAg carrier) or Hepatitis C seropositivity
* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination
* History of seizures
* Febrile or acute illness on the day of inclusion.

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 622 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur Inc.
Locations (2):
- South Africa (2):
  - Soweto, Johannesburg
  - Bertsham

REFERENCES:
- [Result] Madhi SA, Mitha I, Cutland C, Groome M, Santos-Lima E. Immunogenicity and safety of an investigational fully liquid hexavalent combination vaccine versus licensed combination vaccines at 6, 10, and 14 weeks of age in healthy South African infants. Pediatr Infect Dis J. 2011 Apr;30(4):e68-74. doi: 10.1097/INF.0b013e31820b93d2. PMID 21289531
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 28 August 2006 to 11 February 2007 in 2 clinical centers in South Africa.
Pre-assignment Details: A total of 622 of the 715 recruited participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-Hep B-PRP~T Group: Participants received a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular(aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP-T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
- CombAct-Hib™ + Engerix B™ + OPV Group: Participants received a primary series of 3 doses of commercial CombAct-Hib™ vaccine, Engerix B™ vaccine, and oral poliovirus vaccine, with 1 dose of each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
- DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group: Participants received Engerix B™ vaccine at birth, followed by a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular (aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP-T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
Period: Overall Study
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Started | 243 | 242 | 137
Completed | 233 | 235 | 134
Not Completed | 10 | 7 | 3
Not completed — Serious Adverse Event | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 6 | 4 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group | Total
Number analyzed (Participants) | 243 | 242 | 137 | 622
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 243 | 242 | 137 | 622
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 1.04 (0.729) | 1.07 (0.762) | 1.11 (0.773) | 1.07 (0.751)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 118 | 68 | 317
  Male | 112 | 124 | 69 | 305
Region of Enrollment [Number; unit: Participants]
  South Africa | 243 | 242 | 137 | 622

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroprotection After Primary Series Vaccination With DTaP-IPV-Hep B-PRT~T or CombAct Hib™ + Engerix B™ + Oral Polio Vaccine (OPV)
Description: Antibodies were measured by the following methods: anti-Hepatitis B (Hep B) by enhanced chemiluminescence detection, anti-Haemophilus influenzae type b (Hib) by Farr type radio immunoassay, anti-Diphtheria (D) by toxin neutralization assay, anti-Tetanus (T) by indirect enzyme-linked immunosorbent assay (ELISA), and anti-Poliovirus types 1, 2, and 3 by neutralization assay. Seroprotection was defined as the following antibody titers: Anti-Tetanus ≥ 0.01 International Unit (IU)/mL; Anti-Diphtheria ≥ 0.01 IU/mL; Anti-Hepatitis B ≥ 10 mIU/mL; Anti-Polyribosyl ribitol phosphate ≥ 0.15 µg/mL; Anti-polio 1, 2, and 3 ≥ 8 (1/dil).
Time Frame: 1 month post-Dose 3
Population: Seroprotection was assessed in all participants who did not have any protocol violation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 220 | 212 | 123
Participants
  Anti-Hep B (N = 184, 194, 98) | 176 | 185 [0 to 0] | 97 [0 to 0]
  Anti-PRP (N = 219, 212, 122) | 209 | 212 [0 to 0] | 119 [0 to 0]
  Anti-Diphtheria (N = 206, 206, 122) | 201 | 198 [0 to 0] | 116 [0 to 0]
  Anti-Tetanus (N = 213, 210, 122) | 213 | 210 [0 to 0] | 122 [0 to 0]
  Anti-Polio Type 1 (N = 186, 187, 104) | 186 | 174 [0 to 0] | 103 [0 to 0]
  Anti-Polio Type 2 (N = 196, 192, 113) | 193 | 192 [0 to 0] | 111 [0 to 0]
  Anti-Polio Type 3 (N = 182, 179, 98) | 182 | 176 [0 to 0] | 98 [0 to 0]

2. Secondary Outcome: Number of Participants Attaining Other Seroprotection and Seroconversion Titers After Primary Series Vaccination With DTaP-IPV-Hep B-PRT~T (With or Without Engerix B™ at Birth) or CombAct Hib™ + Engerix B™ + Oral Polio Vaccine (OPV)
Description: Anti-Hepatitis B (Hep B) was measured by enhanced chemiluminescence detection, anti-Haemophilus influenzae type b (Hib) by Farr type radio immunoassay, anti diphtheria by toxin neutralization assay, anti-Tetanus (T) by indirect enzyme-linked immunosorbent assay (ELISA), and anti-Pertussis toxoid (PT) and anti-Filamentous hemagglutinin (FHA) by ELISA. Seroprotection was defined as a titer ≥ 100 mIU/mL for anti-Hep B; ≥ 1 µg/mL for anti-PRP; ≥ 0.1 IU/mL (Level 1) and ≥ 1.0 IU/mL (Level 2) for anti-Diphtheria and anti-Tetanus. Seroconversion for anti-PT and anti-FHA was a ≥ 4-fold increase from baseline.
Time Frame: 1 month post-Dose 3
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group: Participants received Engerix B™ vaccine at birth, followed by a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular (aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 220 | 212 | 123
Participants
  Anti-Hep B (N = 184, 194, 98) | 145 | 127 [0 to 0] | 95 [0 to 0]
  Anti-PRP (N = 219, 212, 122) | 174 | 196 [0 to 0] | 97 [0 to 0]
  Anti-Diphtheria Level 1 ( N = 206, 206, 122) | 82 | 28 [0 to 0] | 48 [0 to 0]
  Anti-Diphtheria Level 2 (N = 206, 206, 122) | 3 | 0 [0 to 0] | 4 [0 to 0]
  Anti-Tetanus Level 1 (N = 213, 210, 122) | 213 | 210 [0 to 0] | 122 [0 to 0]
  Anti-Tetanus Level 2 (N = 213, 210, 122) | 158 | 173 [0 to 0] | 83 [0 to 0]
  Anti-Pertussis Toxoid (N = 172, 137, 103) | 161 | 114 [0 to 0] | 98 [0 to 0]
  Anti-FHA (N = 160, 130, 90) | 149 | 75 [0 to 0] | 81 [0 to 0]

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies After Primary Series Vaccination With DTaP-IPV-Hep B-PRT~T (With or Without Engerix B™ at Birth) or CombAct Hib™ + Engerix B™ + Oral Polio Vaccine (OPV)
Description: Anti-Hepatitis B (Hep B) was measured by enhanced chemiluminescence detection, anti-Haemophilus influenzae type b (Hib) by Farr type radio-immunoassay, anti-Diphtheria by toxin neutralization assay, anti-Tetanus by indirect enzyme-linked immunosorbent assay (ELISA), anti-Poliovirus types 1, 2, and 3 by neutralization assay, and anti-Pertussis toxoid (PT) and anti-Filamentous hemagglutinin (FHA) by ELISA.
Time Frame: Day 42 before Dose 1 and 1 month post-Dose 3
Population: GMTs were assessed in all participants who did not have any protocol violation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- DTaP-IPV-Hep B-PRP-T (Engerix B™ at Birth) Group: Participants received Engerix B™ vaccine at birth, followed by a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular (aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP-T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 220 | 212 | 123
Titers
  Anti-Hep B Post-dose 3 (N = 184, 194, 98) | 330 [259 to 420] | 148 [120 to 181] | 1913 [1457 to 2513]
  Anti-PRP Post-dose 3 (N = 219, 212, 122) | 3.31 [2.69 to 4.08] | 5.18 [4.47 to 6.00] | 3.83 [2.92 to 5.02]
  Anti-Diphtheria Post-dose 3 (N = 206, 206, 122) | 0.074 [0.062 to 0.088] | 0.040 [0.035 to 0.046] | 0.074 [0.059 to 0.094]
  Anti-Tetanus Post-dose 3 (N = 213, 210, 122) | 1.51 [1.37 to 1.65] | 1.88 [1.70 to 2.07] | 1.33 [1.17 to 1.51]
  Anti-Polio Type 1 Post-dose 3 (N = 186, 187, 104) | 579 [478 to 702] | 198 [153 to 256] | 557 [410 to 756]
  Anti-Polio Type 2 Post-dose 3 (N = 196, 192, 113) | 620 [512 to 750] | 446 [374 to 533] | 371 [281 to 489]
  Anti-Polio Type 3 Post-dose 3 (N = 182, 179, 98) | 975 [812 to 1170] | 228 [185 to 280] | 811 [645 to 1020]
  Anti-PT Pre-Dose 1 (N = 192, 174, 118) | 7.77 [6.56 to 9.21] | 7.66 [6.23 to 9.42] | 6.62 [5.29 to 8.30]
  Anti-PT Post-dose 3 (N = 192, 156, 108) | 332 [304 to 362] | 191 [147 to 249] | 288 [256 to 323]
  Anti-FHA Pre-dose 1 (N = 192, 175, 107) | 9.27 [8.02 to 10.7] | 8.02 [6.82 to 9.42] | 8.30 [6.80 to 10.1]
  Anti-FHA Post-dose 3 (N = 178, 153, 99) | 207 [190 to 226] | 37.4 [33.4 to 41.9] | 188 [166 to 212]

4. Secondary Outcome: Number of Participants With Antibody Persistence Pre-Booster and Response Post-Booster Vaccination With DTaP-IPV-Hep B-PRT~T (With or Without Engerix B™ at Birth) or CombAct Hib™ + Engerix B™ + OPV
Description: Antibodies were measured by the following methods: anti-Hepatitis B (Hep B) by enhanced chemiluminescence detection, anti-Haemophilus influenzae type b (PRP) by Farr type radio immunoassay, anti-Diphtheria by toxin neutralization assay, anti-Tetanus by indirect enzyme-linked immunosorbent assay (ELISA), anti-poliovirus types 1, 2, and 3 by neutralization assay. Persistence and response were defined as a titer ≥ 10 mIU/mL for anti-Hep B, ≥ 0.15 µg/mL for anti-PRP, ≥ 0.01 IU/mL for anti-Diphtheria and anti-Tetanus, ≥ 8 (1/dil) for anti-Poliovirus, and ≥ 4 EU/mL for anti-PT and anti-FHA.
Time Frame: Day 540 pre-booster and Day 570 post-booster
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- DTaP-IPV-Hep B-PRP-T Group: Participants received a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular(aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP-T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
Arm/Group | DTaP-IPV-Hep B-PRP-T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 204 | 202 | 116
Participants
  Anti-Hep B Pre (N = 199, 199, 113) | 157 | 183 [0 to 0] | 107 [0 to 0]
  Anti-Hep B Post (N = 197, 0, 113) | 194 | 0 [0 to 0] | 113 [0 to 0]
  Anti-PRP Pre (N =2 04, 200, 116) | 166 | 185 [0 to 0] | 88 [0 to 0]
  Anti-PRP Post (N = 203, 201, 115) | 203 | 201 [0 to 0] | 115 [0 to 0]
  Anti-Diphtheria Pre (N = 197, 201, 116) | 184 | 173 [0 to 0] | 98 [0 to 0]
  Anti-Diphtheria Post (N = 195, 200, 111) | 195 | 200 [0 to 0] | 111 [0 to 0]
  Anti-Tetanus Pre (N = 189, 195, 116) | 189 | 195 [0 to 0] | 116 [0 to 0]
  Anti-Tetanus Post (N = 200, 199, 114) | 200 | 199 [0 to 0] | 114 [0 to 0]
  Anti-Polio Type 1 Pre (N = 190, 189, 112) | 185 | 178 [0 to 0] | 108 [0 to 0]
  Anti-Polio Type 1 Post (N = 189, 191, 108) | 189 | 186 [0 to 0] | 108 [0 to 0]
  Anti-Polio Type 2 Pre (N = 190, 191, 111) | 187 | 190 [0 to 0] | 109 [0 to 0]
  Anti-Polio Type 2 Post (N = 191, 190, 107) | 191 | 190 [0 to 0] | 107 [0 to 0]
  Anti-Polio Type 3 Pre (N = 189, 189, 111) | 186 | 185 [0 to 0] | 110 [0 to 0]
  Anti-Polio Type 3 Post (N = 188, 187, 108) | 188 | 185 [0 to 0] | 108 [0 to 0]
  Anti-PT Pre (N = 164, 141, 104) | 151 | 100 [0 to 0] | 95 [0 to 0]
  Anti-PT Post (N= 187, 184, 109) | 187 | 173 [0 to 0] | 109 [0 to 0]
  Anti-PT Post/Pre Ratio (N = 153, 133, 99) | 145 | 111 [0 to 0] | 93 [0 to 0]
  Anti-FHA Pre (N = 173, 148, 103) | 170 | 99 [0 to 0] | 102 [0 to 0]
  Anti-FHA Post (N = 184, 190, 105) | 184 | 190 [0 to 0] | 105 [0 to 0]
  Anti-FHA Post/Pre Ratio (N = 159, 143, 94) | 145 | 138 [0 to 0] | 89 [0 to 0]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Pre- and Post-Booster Vaccination With DTaP-IPV-Hep B-PRT~T (With or Without Engerix B™ at Birth) or CombAct Hib™ + Engerix B™ + OPV
Description: Anti-Hepatitis B (Hep B) was measured by enhanced chemiluminescence detection, anti-Haemophilus influenzae type b (PRP) by Farr type radio immunoassay, anti-Diphtheria by toxin neutralization assay, anti-Tetanus (T) by indirect enzyme-linked immunosorbent assay (ELISA), anti-Poliovirus types 1, 2, and 3 by neutralization assay, and anti-Pertussis toxoid (PT) and anti-Filamentous hemagglutinin (FHA) by ELISA.
Time Frame: Day 540 pre-booster and Day 570, post-booster
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- DTaP-IPV-Hep B-PRP-T Group: Participants received a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular(aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
- DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group: Participants received Engerix B™ vaccine at birth, followed by a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular(aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
Arm/Group | DTaP-IPV-Hep B-PRP-T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 204 | 202 | 116
Titers
  Anti-Hep B Pre (N = 199, 199, 113) | 51.3 [40.0 to 65.8] | 103 [83.3 to 127] | 228 [172 to 303]
  Anti-Hep B Post (N = 197, 0, 113) | 4630 [3402 to 6302] | 0 [0 to 0] | 44893 [33652 to 59890]
  Anti-Hep B Post/Pre Ratio (N = 192, 0, 112) | 88.7 [74.0 to 106] | 0 [0 to 0] | 191 [157 to 231]
  Anti-PRP Pre (N = 204, 200, 116) | 0.757 [0.585 to 0.980] | 1.19 [0.948 to 1.48] | 0.631 [0.448 to 0.889]
  Anti-PRP Post (N = 203, 201, 116) | 68.5 [55.7 to 84.2] | 52.2 [43.9 to 62.2] | 63.1 [47.6 to 83.8]
  Anti-PRP Post/Pre Ratio (N = 203, 199, 115) | 89.0 [71.4 to 111] | 43.6 [34.5 to 55.0] | 97.4 [71.7 to 132]
  Anti-Diphtheria Pre (N = 197, 201, 116) | 0.060 [0.050 to 0.073] | 0.027 [0.023 to 0.032] | 0.045 [0.033 to 0.059]
  Anti-Diphtheria Post (N = 195, 200, 111) | 9.37 [8.05 to 10.9] | 3.33 [2.92 to 3.80] | 7.00 [5.61 to 8.72]
  Anti-Diphtheria Post/Pre Ratio (N = 189, 199, 111) | 158 [137 to 182] | 123 [108 to 140] | 153 [125 to 189]
  Anti-Tetanus Pre (N = 189, 195, 116) | 0.219 [0.189 to 0.254] | 0.311 [0.276 to 0.352] | 0.173 [0.143 to 0.208]
  Anti-Tetanus Post (N = 200, 199, 114) | 10.0 [8.65 to 11.7] | 8.23 [7.49 to 9.04] | 8.13 [6.68 to 9.89]
  Anti-Tetanus Post/Pre Ratio (N = 185, 192, 114) | 45.5 [40.0 to 51.8] | 26.5 [23.5 to 29.9] | 47.4 [39.8 to 56.3]
  Anti-Polio Type 1 Pre (N = 190, 189, 112) | 127 [104 to 155] | 151 [118 to 192] | 142 [107 to 190]
  Anti-Polio Type 1 Post (N = 189, 191, 108) | 7298 [6202 to 8588] | 329 [260 to 417] | 5346 [4309 to 6633]
  Anti-Polio Type 1 Post/Pre Ratio (N=178, 181, 105) | 59.0 [47.0 to 74.0] | 2.27 [1.80 to 2.85] | 38.4 [27.4 to 53.7]
  Anti-Polio Type 2 Pre (N = 190, 191, 111) | 210 [170 to 260] | 246 [204 to 296] | 191 [144 to 255]
  Anti-Polio Type 2 Post (N = 191, 190, 107) | 6637 [5745 to 7668] | 863 [665 to 1118] | 4190 [3460 to 5074]
  Anti-Polio Type 2 Post/Pre Ratio (N=179, 182, 103) | 32.4 [24.9 to 42.3] | 3.82 [2.90 to 5.04] | 23.2 [16.2 to 33.3]
  Anti-Polio Type 3 Pre (N = 189, 189, 111) | 161 [130 to 199] | 114 [96.4 to 135] | 127 [97.9 to 165]
  Anti-Polio Type 3 Post (N = 188, 187, 108) | 6411 [5525 to 7493] | 315 [245 to 404] | 5144 [4156 to 6367]
  Anti-Polio Type 3 Post/Pre Ratio (N=176, 180, 106) | 40.5 [31.0 to 53.0] | 2.92 [2.26 to 3.77] | 41.2 [29.3 to 57.9]
  Anti PT Pre (N=164, 141, 104) | 11.6 [9.88 to 13.6] | 10.4 [8.03 to 13.6] | 12.0 [9.62 to 14.9]
  Anti PT Post (N=187, 184, 109) | 288 [260 to 318] | 110 [88.7 to 137] | 235 [206 to 268]
  Anti-PT Post/Pre Ratio (N=153, 133, 99) | 26.1 [21.8 to 31.1] | 10.6 [8.56 to 13.1] | 20.5 [16.5 to 25.4]
  Anti-FHA Pre (N = 173, 148, 103) | 30.5 [25.4 to 36.7] | 5.43 [4.52 to 6.53] | 25.1 [19.7 to 31.9]
  Anti-FHA Post (N = 184, 190, 105) | 570 [514 to 630] | 211 [193 to 231] | 472 [419 to 533]
  Anti-FHA Post/Pre Ratio (N = 159, 143, 94) | 18.9 [15.8 to 22.6] | 40.8 [34.5 to 48.1] | 20.3 [16.5 to 24.9]

6. Secondary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactions After Primary Vaccination Series With With DTaP-IPV-Hep B-PRT~T (With or Without Engerix B™ at Birth) or CombAct Hib™ + Engerix B™ + Oral Polio Vaccine (OPV).
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited System Reactions: Fever (Temperature), Vomiting, Crying, Somnolence, Anorexia, Irritability. Grade 3 was defined as: Pain - crying when injected limb is moved or the movement reduced; Erythema and Swelling - ≥ 5 cm; Fever - temperature ≥ 39.0ºC; Vomiting - ≥ 6 episodes/24 hours or requiring parenteral hydration; Crying abnormal - > 3 hours; Somnolence - sleeping most of the time or difficulty to wake up; Anorexia - refusing ≥ 3 feeds or refusing most feeds/meals; and Irritability - inconsolable.
Time Frame: Day 0 up to Day 7 post each dose
Population: Solicited reactions were assessed in all participants who received at least 1 dose of investigational or reference vaccine, according to the vaccine actually received - Safety Analysis Population.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 243 | 242 | 137
Participants
  Pain Post-dose 1 (N = 234, 237, 134) | 166 | 177 [0 to 0] | 95 [0 to 0]
  Pain Post-dose 2 (N = 234, 233, 134) | 171 | 171 [0 to 0] | 97 [0 to 0]
  Pain Post-dose 3 ( N = 232, 234, 134) | 143 | 162 [0 to 0] | 83 [0 to 0]
  Grade 3 Pain Post-Any Dose (N = 237, 238, 136) | 17 | 24 [0 to 0] | 7 [0 to 0]
  Erythema Post-dose 1 (N = 233, 237, 132) | 112 | 133 [0 to 0] | 69 [0 to 0]
  Erythema Post-dose 2 (N = 232, 231, 133) | 116 | 114 [0 to 0] | 59 [0 to 0]
  Erythema Post-dose 3 (N = 231, 234, 132) | 103 | 106 [0 to 0] | 56 [0 to 0]
  Grade 3 Erythema Post-Any Dose (N = 236, 238, 135) | 9 | 15 [0 to 0] | 2 [0 to 0]
  Swelling Post-dose 1 (N = 231, 238, 134) | 87 | 102 [0 to 0] | 48 [0 to 0]
  Swelling Post-dose 2 (N = 233, 230, 133) | 88 | 109 [0 to 0] | 43 [0 to 0]
  Swelling Post-dose 3 (N = 232, 232, 133) | 74 | 89 [0 to 0] | 39 [0 to 0]
  Grade 3 Swelling Post-Any Dose (N = 236, 238, 136) | 9 | 10 [0 to 0] | 4 [0 to 0]
  Pyrexia Post-dose 1 (N = 234, 238, 132) | 50 | 38 [0 to 0] | 27 [0 to 0]
  Pyrexia Post-dose 2 (N = 234, 232, 134) | 43 | 35 [0 to 0] | 18 [0 to 0]
  Pyrexia Post-dose 3 (N = 230, 232, 134) | 48 | 34 [0 to 0] | 21 [0 to 0]
  Grade 3 Pyrexia Post-Any Dose (N = 236, 238, 136) | 4 | 1 [0 to 0] | 0 [0 to 0]
  Vomiting Post-dose 1 (N = 233, 238, 133) | 59 | 59 [0 to 0] | 30 [0 to 0]
  Vomiting Post-dose 2 (N = 234, 233, 134) | 52 | 56 [0 to 0] | 35 [0 to 0]
  Vomiting Post-dose 3 (N = 231, 233, 134) | 56 | 49 [0 to 0] | 31 [0 to 0]
  Grade 3 Vomiting Post-Any Dose (N = 236, 238, 135) | 14 | 7 [0 to 0] | 6 [0 to 0]
  Crying Post-dose 1 (N = 234, 238, 133) | 138 | 154 [0 to 0] | 91 [0 to 0]
  Crying Post-dose 2 (N = 234, 233, 134) | 131 | 135 [0 to 0] | 74 [0 to 0]
  Crying Post-dose 3 (N = 231, 233, 134) | 106 | 116 [0 to 0] | 66 [0 to 0]
  Grade 3 Crying Post-Any Dose (N = 236, 238, 135) | 15 | 20 [0 to 0] | 9 [0 to 0]
  Somnolence Post-dose 1 (N = 232, 238, 133) | 100 | 103 [0 to 0] | 57 [0 to 0]
  Somnolence Post-dose 2 (N = 234, 232, 134) | 79 | 90 [0 to 0] | 47 [0 to 0]
  Somnolence Post-dose 3 (N = 231, 232, 134) | 72 | 69 [0 to 0] | 43 [0 to 0]
  Grade 3 Somnolence Post-Any Dose (N=236, 238, 135) | 9 | 9 [0 to 0] | 8 [0 to 0]
  Anorexia Post-dose 1 (N = 233, 238, 134) | 62 | 87 [0 to 0] | 42 [0 to 0]
  Anorexia Post-dose 2 (N = 234, 232, 134) | 66 | 68 [0 to 0] | 39 [0 to 0]
  Anorexia Post-dose 3 (N = 231, 232, 134) | 64 | 76 [0 to 0] | 39 [0 to 0]
  Grade 3 Anorexia Post-Any Dose (N=236, 238, 136) | 9 | 13 [0 to 0] | 5 [0 to 0]
  Irritability Post-dose 1 (N=234, 238, 132) | 128 | 137 [0 to 0] | 77 [0 to 0]
  Irritability Post-dose 2 (N = 234, 232, 134) | 114 | 118 [0 to 0] | 66 [0 to 0]
  Irritability Post-dose 3 (N = 231, 232, 134) | 94 | 99 [0 to 0] | 53 [0 to 0]
  Grd 3 Irritability Post-Any Dose (N=236, 238, 135) | 18 | 16 [0 to 0] | 5 [0 to 0]

7. Secondary Outcome: Number of Participants With Solicited Injection Site (Study Vaccine Site) and Systemic Reactions After Booster Vaccination With DTaP-IPV-Hep B-PRT~T (With or Without Engerix B™ at Birth) or CombAct Hib™ + Engerix B™ + Oral Polio Vaccine (OPV)
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling, and Extensive swelling of vaccinated limb. Solicited System Reactions: Fever (Temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability. Grade 3 was defined as: Pain, crying when injected limb is moved or the movement reduced; Erythema and Swelling, ≥ 5 cm; Fever, temperature ≥ 39.0ºC; Vomiting, ≥ 6 episodes/24 hours or requiring parenteral hydration; Crying, > 3 hours; Somnolence, sleeping most of the time or difficulty to wake up; Anorexia, refusing ≥ 3 feeds or refusing most feeds/meals; and Irritability, inconsolable.
Time Frame: Day 0 up to 7 post-booster vaccination
Population: Solicited reactions were assessed in all participants who received at least 1 dose of investigational or reference vaccine, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Participants
Groups:
- DTaP-IPV-Hep B-PRP~T Group: Participants received a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular(aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
- DTaP-IPV-Hep B-PRP-T (Engerix B™ at Birth) Group: Participants received Engerix B™ vaccine at birth, followed by a primary series of 3 doses of diphtheria (D), tetanus (T), pertussis (2 component acellular(aP), recombinant hepatitis B Hansenula (Hep B) and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate (PRP) conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with 1 dose each at 6, 10, and 14 weeks of age, and a booster dose at 15 to 18 months of age. Participants also received Trimovax™ and Varilrix™ vaccines at 15 to 18 months of age.
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP-T (Engerix B™ at Birth) Group
Number analyzed (Participants) | 218 | 219 | 130
Participants
  Pain | 138 | 149 [0 to 0] | 84 [0 to 0]
  Grade 3 Pain | 5 | 4 [0 to 0] | 1 [0 to 0]
  Erythema | 102 | 104 [0 to 0] | 54 [0 to 0]
  Grade 3 Erythema | 3 | 2 [0 to 0] | 2 [0 to 0]
  Swelling | 75 | 98 [0 to 0] | 48 [0 to 0]
  Grade 3 Swelling | 2 | 11 [0 to 0] | 5 [0 to 0]
  Extensive swelling of vaccinated limb | 0 | 0 | 0
  Grade 3 Extensive swelling of vaccinated limb | 0 | 0 | 0
  Pyrexia | 61 | 50 [0 to 0] | 37 [0 to 0]
  Grade 3 Pyrexia | 1 | 2 [0 to 0] | 2 [0 to 0]
  Vomiting | 22 | 28 [0 to 0] | 14 [0 to 0]
  Grade 3 Vomiting | 0 | 2 [0 to 0] | 0 [0 to 0]
  Crying | 106 | 115 [0 to 0] | 58 [0 to 0]
  Grade 3 Crying | 3 | 0 [0 to 0] | 2 [0 to 0]
  Somnolence | 85 | 80 [0 to 0] | 43 [0 to 0]
  Grade 3 Somnolence | 3 | 1 [0 to 0] | 1 [0 to 0]
  Anorexia | 88 | 99 [0 to 0] | 55 [0 to 0]
  Grade 3 Anorexia | 8 | 4 [0 to 0] | 4 [0 to 0]
  Irritability | 98 | 103 [0 to 0] | 52 [0 to 0]
  Grade 3 Irritability | 2 | 1 [0 to 0] | 1 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the time of each vaccination up to 28 days after each primary and the booster vaccination.
Description: The total number of participants for which safety data were collected following booster vaccination were less than those for the primary vaccination. The total number for each event represents participants that were available for the data or endpoint.
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | CombAct-Hib™ + Engerix B™ + OPV Group | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group
Serious Adverse Events (participants affected / at risk) | 7/243 | 6/242 | 5/137
Other Adverse Events (participants affected / at risk) | 202/243 | 210/242 | 119/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T Group (N=243) | CombAct-Hib™ + Engerix B™ + OPV Group (N=242) | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group (N=137)
Pulmonary Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Disease Congenital (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Dysentery (Infections and infestations) | 0/218 (0) | 0 (0) | 1/130 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1/130 (1)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0)
Failure to Thrive (Metabolism and nutrition disorders) | 1/218 (1) | 0/219 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T Group (N=243) | CombAct-Hib™ + Engerix B™ + OPV Group (N=242) | DTaP-IPV-Hep B-PRP~T (Engerix B™ at Birth) Group (N=137)
Vomiting (Gastrointestinal disorders) | 106/236 (106) | 100/238 (100) | 54/135 (54)
Injection Site Bruising (General disorders) | 6/237 (6) | 9/238 (9) | 9/136 (9)
Injection Site Pain (General disorders) | 202/237 (202) | 210/238 (210) | 119/136 (119)
Injection Site Erythema (General disorders) | 160/236 (160) | 173/238 (173) | 91/135 (91)
Injection Site Swelling (General disorders) | 130/236 (130) | 150/238 (150) | 65/136 (65)
Irritability (General disorders) | 157/236 (157) | 165/238 (165) | 94/135 (94)
Pyrexia (General disorders) | 105/236 (105) | 79/238 (79) | 45/136 (45)
Upper Respiratory Tract Infection (Infections and infestations) | 11/237 (11) | 13/238 (13) | 4/136 (4)
Anorexia (Metabolism and nutrition disorders) | 110/236 (110) | 133/238 (133) | 67/136 (67)
Somnolence (Nervous system disorders) | 143/236 (143) | 143/238 (143) | 78/135 (78)
Crying (Psychiatric disorders) | 180/236 (180) | 186/238 (186) | 112/135 (112)
Cough (Respiratory, thoracic and mediastinal disorders) | 13/237 (13) | 4/238 (4) | 4/136 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications